CLINICAL TRIAL: NCT03040570
Title: A Randomised Pilot Multiple Centre Trial of Conservative Versus Liberal Oxygenation Targets in Critically Ill Children
Brief Title: Conservative Versus Liberal Oxygenation Targets in Critically Ill Children
Acronym: Oxy-PICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Intensive Care National Audit & Research Centre (Other); University of Southampton (Other); St Mary's Hospital, London (Other); University Hospital Southampton NHS Foundation Trust (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15IA35
Record Dates: First submitted 2016-11-21; First posted 2017-02-02 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Critical Care; Hypoxia; Pediatric ALL
MeSH Terms: conditions — Hypoxia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative oxygenation target (Experimental): Children in the conservative oxygenation target group receive treatment targeting oxygen saturation values of 88-92%.
  Interventions: Procedure: Conservative oxygenation target
- Liberal oxygenation target (Active Comparator): Children in the liberal oxygenation target group receive treatment targeting oxygen saturation values of >94%.
  Interventions: Procedure: Liberal oxygenation target

INTERVENTIONS:
Procedure: Conservative oxygenation target — Participants allocated to the conservative oxygenation target group will receive supplemental oxygen and ventilator settings at the discretion of the treating clinical team with the aim of peripheral oxygen saturations remaining 88-92% (inclusive).
  Arms: Conservative oxygenation target
Procedure: Liberal oxygenation target — Participants allocated to the liberal oxygenation target group will receive supplemental oxygen and ventilator settings at the discretion of the treating clinical team with the aim of peripheral oxygen saturations remaining >94%.
  Arms: Liberal oxygenation target

SUMMARY:
A feasibility study to determine if it is possible to perform a safe, adequately powered, and affordable multi-centre study in critically ill children comparing current practice of liberal targets for systemic oxygen levels with more conservative targets.

DETAILED DESCRIPTION:
Around 19,000 critically ill children are admitted to paediatric intensive care units (PICU) each year in the UK. A large number of these children need breathing support, and this is usually provided through an invasive machine called a 'ventilator'. Clinicians make decisions for treatment based on how much oxygen their patient has in their blood (this is called oxygen saturation or oxygenation) and currently the amount of oxygen critically ill children need is not fully understood. This means that some clinicians use a lower oxygen saturation target, and others, a higher target. This may be problematic as research in neonates (babies) and adults has shown that oxygen saturation levels can influence a patient's chance of survival, how long they stay in hospital and healthcare costs.

Response to oxygen is different in babies, children and adults. This means that the results from the neonatal and adult research are unlikely to be valid or applicable in children due to age-related differences. Urgent high quality clinical evidence is therefore needed to inform on the best targets of oxygenation during critical illness in children.

As large clinical trials are expensive to conduct, it is important to demonstrate that a large-scale trial can be done and that the different components of a trial can all work together. Therefore, the Oxy-PICU study is a 'pilot randomised clinical trial' (a smaller version of the trial we would like to conduct) and will test the feasibility and safety of conducting a large scale trial comparing a restrictive oxygen saturation target (88-92%) with a more liberal oxygen saturation target (>94%). Oxy-PICU will also collect blood and urine samples to allow for in depth study of the biology of the different oxygenation targets.

The pilot trial will take place at three PICUs (two in London and one in Southampton) and aims to include between 115-125 eligible children over six months. Given the emergency nature of these children and the need to provide immediate care, informed consent will be sought after the children are entered into the study (this is known as deferred consent).

ELIGIBILITY:
Inclusion Criteria:

* less than 16 years and > 38 weeks corrected gestational age
* receiving supplemental oxygen for abnormal gas exchange
* emergency admission accepted to a participating paediatric intensive care unit (PICU) requiring mechanical ventilation within first 6 hours of face-to-face contact with PICU staff or transport team

Exclusion Criteria:

* recruited to Oxy-PICU in a previous admission
* brain pathology/injury as a primary reason for admission (e.g traumatic brain injury, post-cardiac arrest, stroke, convulsive status epilepticus without aspiration)
* known pulmonary hypertension
* known or suspected sickle cell disease
* known or suspected uncorrected congenital cardiac disease
* End-of-life care plan in place with limitation of resuscitation
* not expected to survive PICU admission
* receiving long-term mechanical ventilation prior to this admission (non-invasive ventilation or invasive ventilation)

Ages: 39 Weeks to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Number of eligible patients recruited per site per month | Baseline

SECONDARY OUTCOMES:
Proportion of parents/legal representatives refusing deferred consent | Through study completion, an average of 24 hours
Proportion of eligible patients randomised | Baseline
Distribution of time to randomisation | Baseline
Proportion of systemic oxygen saturations within the target range in each group | Through study completion, an average of 72 hours
Proportion of patients in each arm requiring other treatments influencing tissue oxygen delivery (blood transfusion, inotropic support) | Through study completion, an average of 72 hours
Length of ventilation - proportion of randomised patients with outcome available in each group | Through study completion, an average of 2 days
Length of ventilation - mean (standard deviation) in each group | Through study completion, an average of 2 days
Length of ventilation - median and quartiles in each group. | Through study completion, an average of 2 days
Observed adverse events | 28 days
Time taken for data collection and entry | 28 days
Measurement of ischemia-modified albumin (plasma) | 72 hours
Measurement of malondialdehyde (plasma) | 72 hours
Measurement of total antioxidant status (plasma) | 72 hours
Length of PICU stay - proportion of randomised patients with outcome available in each group | Through study completion, an average of 2 days
Length of PICU stay - mean (standard deviation) in each group. | Through study completion, an average of 2 days
Length of PICU stay - median and quartiles in each group. | Through study completion, an average of 2 days
Hospital mortality - proportion of randomised patients with outcome available in each group | Through study completion, an average of 2 days
Hospital mortality - number (percentage) in each group. | Through study completion, an average of 2 days
PICU mortality - proportion of randomised patients with outcome available in each group | Through study completion, an average of 2 days
PICU mortality - number (percentage) in each group. | Through study completion, an average of 2 days
Days of organ specific support - proportion of randomised patients with outcome available in each group | Through study completion, an average of 2 days
Days of organ specific support - mean (standard deviation) in each group | Through study completion, an average of 2 days
Days of organ specific support - median and quartiles in each group | Through study completion, an average of 2 days
Measurement of hypoxia-inducible factor-1 alpha mRNA expression (leukocytes) | 72 hours

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Great Ormond Street Hospital for Children, London
  - St Mary's Hospital, London
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Jones GAL, Eaton S, Orford M, Ray S, Wiley D, Ramnarayan P, Inwald D, Grocott MPW, Griksaitis M, Pappachan J, O'Neill L, Mouncey PR, Harrison DA, Rowan KM, Peters MJ; Oxy-PICU Investigators of the Paediatric Critical Care Society Study Group (PCCS-SG). Randomization to a Liberal Versus Conservative Oxygenation Target: Redox Responses in Critically Ill Children. Pediatr Crit Care Med. 2023 Mar 1;24(3):e137-e146. doi: 10.1097/PCC.0000000000003175. Epub 2023 Jan 19. PMID 36728001
- [Derived] Peters MJ, Jones GAL, Wiley D, Wulff J, Ramnarayan P, Ray S, Inwald D, Grocott M, Griksaitis M, Pappachan J, O'Neill L, Eaton S, Mouncey PR, Harrison DA, Rowan KM; Oxy-PICU Investigators for the Paediatric Intensive Care Society Study Group (PICS-SG). Conservative versus liberal oxygenation targets in critically ill children: the randomised multiple-centre pilot Oxy-PICU trial. Intensive Care Med. 2018 Aug;44(8):1240-1248. doi: 10.1007/s00134-018-5232-7. Epub 2018 Jun 4. PMID 29868973
- [Derived] Jones GAL, Ramnarayan P, Raman S, Inwald D, Grocott MPW, Eaton S, Ray S, Griksaitis MJ, Pappachan J, Wiley D, Mouncey PR, Wulff J, Harrison DA, Rowan KM, Peters MJ; Oxy-PICU Investigators for thePaediatric Intensive Care Society-Study Group (PICS-SG). Protocol for a randomised pilot multiple centre trial of conservative versus liberal oxygenation targets in critically ill children (Oxy-PICU). BMJ Open. 2017 Dec 14;7(12):e019253. doi: 10.1136/bmjopen-2017-019253. PMID 29247112